CLINICAL TRIAL: NCT03754322
Title: "LAMPREG TRIAL" Active Case Detection and Treatment of Malaria in Pregnancy Using LAMP Technology: A Pragmatic Randomized Multi-Center Diagnostic Outcomes Trial
Brief Title: LAMP Detection of Malaria in PREGnancy (LAMPREG) Trial
Acronym: LAMPREG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Jimma University (Other); Amhara Public Health Institute, Ethiopia (Unknown); Armauer Hansen Research Institute, Ethiopia (Other)
Responsible Party: Principal Investigator, Dylan R Pillai, Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: REB17-1335
Record Dates: First submitted 2018-08-24; First posted 2018-11-27 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Malaria; Pregnancy Malaria; Malaria in Pregnancy
Keywords: Plasmodium; Pregnancy; Malaria; LAMP; Asymptomatic infections; Low Birth Weight; Outcomes
MeSH Terms: conditions — Malaria; Asymptomatic Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (Active Comparator): One third of individuals get allocated to the standard of care arm. At each antenatal visit as per Ethiopian guidelines, pregnant women enrolled in the study will be submitted to the standard of care for malaria in pregnancy. If the pregnant mothers are symptomatic for malaria, they receive microscopy (blood smear for Plasmodium detection) and then are treated with anti-malarial therapy if microscopy is positive for Plasmodium. If it is negative they receive no treatment. If they are asymptomatic, they do not receive any further investigations or treatment in relation to malaria.
  Interventions: Diagnostic Test: Microscopy/RDT
- Intervention arm (Experimental): The remaining two-thirds of participants will be actively screened (symptomatic and asymptomatic) for Plasmodium infection at each antenatal visit, using both LAMP and conventional techniques (microscopy and RDT). If either is positive, participants will be treated with antimalarial therapy according to Ethiopian Ministry of Health guidelines. If both are negative then they receive no treatment.
  Interventions: Diagnostic Test: LAMP; Diagnostic Test: Microscopy/RDT

INTERVENTIONS:
Diagnostic Test: LAMP — LAMP testing involves taking a blood specimen using venous puncture, extracting DNA and performing a commercial CE-marked LAMP malaria assay to obtain a malaria result (presence/absence of parasite DNA) at the species level
  Arms: Intervention arm
Diagnostic Test: Microscopy/RDT — Standard of care management of malaria in pregnancy relies on microscopy and/or RDT for diagnosis

SUMMARY:
Objective: The aim of this study is to evaluate the impact of enhanced malaria cases detection using molecular testing (LAMP) on maternal and infant morbidity and mortality in a prospective study design.

A pragmatic randomized control diagnostic trial will be conducted from October 2020 until March 1 2022 in pregnant mothers at sites in Ethiopia. Both symptomatic and asymptomatic first and early second trimester pregnant women will be included in the study and individually randomized to either standard of care or enhanced cased detection arms using LAMP for malaria. Women (n=2583) will be enrolled during a seven-month period encompassing the peak transmission seasons and then followed until delivery. In the standard of care arm, venous blood sample will be collected from each study participant and the presence of Plasmodium infection will be diagnosed by microscopy in symptomatic patients. Pregnant women who test positive for malaria will be referred and treated for malaria with quinine or artemisinin combination therapies (ACTs) as per national guidelines. In the intervention arm, mothers who are symptomatic or asymptomatic will be tested by a commercially available CE-approved LAMP malaria test and microscopy/RDT for malaria at each clinic visit and treated if positive by any test. Pregnant mothers who require treatment will be referred and treated with either quinine or artemisinin combination therapy (ACTs) as per national guidelines. The primary outcome is the proportion of deliveries with low birth weight based on WHO definition, with secondary outcomes of:(i)absolute birth weight; (ii) maternal hemoglobin;(ii) neonatal hemoglobin at birth;(iv) neonatal mortality; (v) stillbirth; and (vi) prematurity in each arm of the study.

DETAILED DESCRIPTION:
Malaria in pregnancy often results in high degree of morbidity and mortality of the pregnant mother and the fetus. Early and accurate diagnosis of subclinical infections will be critical to malaria elimination and specifically the goals of the World Health Organization to reduce the burden of disease by 90% before 2030. This goal can only be achieved using highly sensitive methods such as LAMP that are capable of detecting subclinical infections with very low parasitemia. Currently both Giemsa stained blood film microscopy and RDT are the only laboratory methods that are used to diagnose malaria both in pregnant mothers and the general population. This leaves a big gap in the detection of low-level infections and asymptomatic malaria due to the documented lack of sensitivity of the aforementioned methods. This, in turn, predisposes pregnant mothers to malaria-related complications that endangers the life of the mother and the fetus. In this study, we propose that the use of a highly sensitive LAMP technique will enable us to detect more asymptomatic Plasmodium infections in pregnant women. This consequently results in early treatment of the pregnant mothers and may avert maternal and fetal morbidity and mortality. This study is of particular importance in Ethiopia where IPT is not used for pregnant women and therefore accurate screening is paramount.

OBJECTIVES

General objective To assess the impact of LAMP in the diagnosis of malaria in pregnancy and its potential role in reducing mortality and morbidity attributable to malaria. We hypothesize that the additional sensitivity of LAMP coupled with active case detection in detecting malaria in pregnancy will result in additional cases being identified and treated.

Specific objectives

1. To evaluate the impact of LAMP versus microscopy/RDT for the detection of malaria in pregnant mothers in terms maternal and infant morbidity and mortality.
2. To evaluate the impact of enhanced case detection of malaria in pregnancy by screening asymptomatic mothers at each antenatal visit until delivery.
3. To determine the impact of treating LAMP-positive asymptomatic and symptomatic pregnant women as compared to standard of care. Treatment is per national guidelines.

MATERIALS AND METHODS

Study area The study will be conducted at sites across several sites in Ethiopia to obtain sufficient enrolment and spanning different transmission settings based on epidemiological data provided by the Federal Ministry of Health. The study sites are in the Amhara region (Chisabay Health center, Hamusit health center and Andasa Health center), and in the Jimma area (Bonga (GebreTsadik Shawo) General hospital, Uffa health center and Lare health center). In Ethiopia, malaria is characterized by its seasonality where the peak transmission season is from October to December with a second peak in June. P. falciparum and P. vivax are the predominant species in the area.

Study design and period

The study is a prospective diagnostic study of malaria in pregnant women. The goal is to determine whether: (i) LAMP provides a clinically measurable benefit compared to current first line diagnostic test of Giemsa-stained microscopy and whether (ii) enhanced case detection of asymptomatic mothers with LAMP has added value in terms of outcomes. We hypothesize that addition of LAMP to one arm will be of greater benefit than microscopy alone due to additional LAMP sensitivity. We further hypothesize that enhanced case detection by screening asymptomatic mothers at each antenatal visit will be of additional value in treating malaria. Both symptomatic and asymptomatic first and second trimester mothers will be included in the study and individually randomized to one of two arms: standard of care or enhanced cased detection arms using LAMP for malaria. Mothers will be enrolled during a seven-month period from June 2021 to January 2022 and then followed until 28 days after delivery. Given the rate of pregnant mothers at the locations, we anticipate that the required minimum of 2583 mothers will be enrolled in the study during the study period. In the first standard of care arm, venous blood sample will be collected from each study participant and the presence of Plasmodium infection will be diagnosed by microscopy in symptomatic patients. Pregnant women who test positive for malaria will be referred and treated for malaria with quinine or ACTs as per national guidelines. In the second (test) arm, mothers whether symptomatic or asymptomatic will be tested by a commercially available CE-approved LAMP malaria test (Human Diagnostics LoopAMP (Wiesbaden, Germany)) at each clinic visit in addition to RDT/microscopy. The commercial LAMP tests can distinguish P. falciparum and P. vivax and treatment will be given according to national guidelines. The purpose of doing all tests in the intervention arm is to determine how many additional cases LAMP identified. The primary outcome is the proportion of deliveries with low birth weight, with secondary outcomes of: (i) absolute birth weight; (ii) maternal hemoglobin; (ii) neonatal hemoglobin at birth (Standard Hgb testing from peripheral blood or finger prick); (iv) neonatal mortality; (v) pregnancy loss; and (vi) prematurity in each of the two arms.

ELIGIBILITY:
Inclusion Criteria:

* Must be a pregnant woman in the first or second trimester at time of enrollment
* Consent to the study

Exclusion Criteria:

* Pregnant woman in the third trimester at time of enrollment
* Multiparity
* Severe malaria at inclusion as per WHO criteria
* At risk pregnancy as per Ethiopian guidelines
* Impossibility to date pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women only
Enrollment: 2424 (Actual)
Dates: Start 2021-06-18 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
Proportion of deliveries with low birth weight | At the head to toe assessment of the baby within 24 hours of delivery
  Birth weight will be considered as low if < 2500 g

SECONDARY OUTCOMES:
Absolute birth weight | At the head to toe assessment of the baby within 24 hours of delivery
  Birth weight in grams
Maternal hemoglobin | During the pregnancy and at delivery
  Maternal hemoglobin in g/dL
Neonatal hemoglobin at birth | At the head to toe assessment of the baby within 24 hours of delivery
  Foetal hemoglobin in g/dL
Proportion of fetal loss | During the study time, for each inclusion until delivery
  Early stillbirth < 20-27 completed weeks of pregnancy Late stillbirth 28 -36 weeks of pregnancy Term still birth > 37 weeks of pregnancy
Prematurity | At delivery
  Baby born Extremely preterm < 28 weeks of pregnancy Very preterm 28-32 weeks of pregnancy Moderate to late preterm 32-37 weeks of pregnancy

OTHER OUTCOMES:
Performance of diagnosis methods compared to qRT-PCR as a gold standard | At the end of the study
  Evaluation of the sensitivity, specificity, PPV and NPV for LAMP, RDT and microscopy in the study
Assessment of the development of placental malaria | At delivery and post hoc
  Evaluation of the presence of malaria pigment in macrophages from placental blood. qPCR in placenta blood

CONTACTS AND LOCATIONS:
Overall Officials: Dylan Pillai, MD, PhD, Principal Investigator — University of Calgary
Locations (4):
- University of Calgary, Calgary, Alberta, Canada
- Ethiopia (3):
  - Amhara Public Health Institute, Bahir Dar, Amhara
  - Tropical & Infectious Diseases Research Center (TIDRC), Jimma University, Jimma, Oromiya
  - Armauer Hansen Research Institute, Ethiopia, Addis Ababa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gebresenbet RF, Kamaliddin C, Bekele ZM, Teferi M, Tegegne B, Yewhalaw D, Bayih AG, Pillai DR; LAMPREG Study Group. Active case detection and treatment of malaria in pregnancy using LAMP technology (LAMPREG): a pragmatic randomised diagnostic outcomes trial-study protocol. BMJ Open. 2022 Jul 18;12(7):e058397. doi: 10.1136/bmjopen-2021-058397. PMID 35851027

DOCUMENTS (2):
  • Study Protocol (2020-03-29): https://cdn.clinicaltrials.gov/large-docs/22/NCT03754322/Prot_002.pdf
  • Statistical Analysis Plan (2021-02-22): https://cdn.clinicaltrials.gov/large-docs/22/NCT03754322/SAP_003.pdf